CLINICAL TRIAL: NCT04093817
Title: Arrhythmia in on Pump vs. Off Pump Coronary Artery Bypass Grafting
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Emad Kamel, resident doctor at cardiothoracic surgery department at Assiut university hospital, Assiut University
Other Study IDs: Arrhythmia in CABG
Record Dates: First submitted 2019-09-06; First posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- on pump CABG: patients under going CABG with cardiopulmonary bypass machine
  Interventions: Device: cardio pulmonary bypass machine
- off pump CABG: patients under going CABG without cardiopulmonary bypass machine

INTERVENTIONS:
Device: cardio pulmonary bypass machine — cardio pulmonary bypass machine is a machine that work to compensate for the function of the heart and the lungs in the operation
  Groups: on pump CABG

SUMMARY:
The aim of this research is to know the incidence of arrhythmias in on vs. off pump CABG and to know their relations to the patient's morbidity and mortality, hospital stay and hospital costs.

DETAILED DESCRIPTION:
On pump vs. off pump CABG has been a topic of debate for many years regarding the benefits and the risks of each technique .Off pump CABG began 30 years ago. Its promotion was based on its potential benefits over some of the limitation of traditional on pump CABG. It avoids the trauma of cardiopulmonary bypass (CPB) and minimizing aortic manipulation and reducing length of hospital stay and morbidity.

There is a criticism regarding completence of revascularization in off pump vs. on pump CABG, this is no longer valid in the current era as technology to safely perform multi vessel off pump has improved tremendously over the past decade.

One of the debates between these two techniques was the incidence of arrhythmias in and after the operation and its relation to morbidity and mortality at the operation and hospital stay after the operation.

As known atrial fibrillation (AF) is still the most common arrhythmia that occur after CABG and although in some studies it has been considered a benign and self-limiting complication, some suggest serious morbidity and mortality from this complication, it is said that it affects more than 40% of patients underwent CABG. Atrial fibrillation (AF) may lead to thromboembolic complications, additional pharmacotherapy, longer hospital stay, increase cost, anxiety and stroke.

Most AF post CABG are found in the second to third post-operative day. SO, on this study the investigators focus one the incidence of arrhythmias, especially AF in those two techniques and their relations to patients' morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* All patients subjected to CABG

Exclusion Criteria:

* Associated valvular heart disease
* Emergency cases
* Previous AF

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients under going coronary artery bypass grafting from ischemic heart disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
the incidence of arrhythmias in on pump vs. off pump coronary artery bypass grafting | the number of episodes of arrhythmia s in one week after the operation
  the frequency of arrhythmia s (in number of episodes) using a12-leads continuous electrocardiogram(ECG) in each type of the two operations.the number of patients that experience those arrhythmia s (in percentage) from the total number of patients that go for those two operations.

SECONDARY OUTCOMES:
decrease morbidity, mortality, hospital stay and hospital cost | baseline
  1. To know the relation of the arrythmias in the number of days that the patient stays after the operation.
  2. To know the relation of the arrhythmias as a cause to the mortality of these patients.(number of patients die after the operation from the total deaths from these two operations).
  3. To know the the relation of the arrhythmias in these two operations to their patients morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Samy Othman, prof.dr, Study Chair — Assiut University; Ahmed Taha, lecturer, Study Chair — Assiut University

REFERENCES:
- [Background] Gaudino M, Angelini GD, Antoniades C, Bakaeen F, Benedetto U, Calafiore AM, Di Franco A, Di Mauro M, Fremes SE, Girardi LN, Glineur D, Grau J, He GW, Patrono C, Puskas JD, Ruel M, Schwann TA, Tam DY, Tatoulis J, Tranbaugh R, Vallely M, Zenati MA, Mack M, Taggart DP; Arterial Grafting International Consortium (ATLANTIC) Alliance. Off-Pump Coronary Artery Bypass Grafting: 30 Years of Debate. J Am Heart Assoc. 2018 Aug 21;7(16):e009934. doi: 10.1161/JAHA.118.009934. No abstract available. PMID 30369328
- [Background] Davoodi S, Karimi A, Ahmadi SH, Marzban M, Movahhedi N, Abbasi K, Omran AS, Shirzad M, Sheikhvatan M, Abbasi SH, Bina P. Early outcome of off-pump versus on-pump coronary revascularization. Pan Afr Med J. 2014 Apr 22;17:309. doi: 10.11604/pamj.2014.17.309.1723. eCollection 2014. PMID 25328605
- [Background] Lewicki L, Siebert J, Rogowski J. Atrial fibrillation following off-pump versus on-pump coronary artery bypass grafting: Incidence and risk factors. Cardiol J. 2016;23(5):518-523. doi: 10.5603/CJ.a2016.0066. Epub 2016 Sep 26. PMID 27665857